CLINICAL TRIAL: NCT04494555
Title: Do Adaptable Sockets Improve Military Performance?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Collaborators: University of Washington (Other)
Responsible Party: Principal Investigator, Dr. Walter Lee Childers, Principle Investigator, Brooke Army Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BAMC C.2020.007
Record Dates: First submitted 2020-05-15; First posted 2020-07-31 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Amputation Stump
Keywords: amputation; bioimpedance; prosthetic socket; transtibial

STUDY DESIGN:
Intervention Model Description: This is a repeated measures prospective study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adaptable Prosthetic Socket (Experimental): Using measurements of limb-socket displacements from sensors embedded within the socket wall, adaptable sockets make small adjustments to socket size so as to maintain consistent displacements while prosthesis users are active. They do not require the user to stop activity or to touch or modify the prosthesis, and they do not distract users from their objectives.
  Interventions: Device: Static socket; Device: User adjusted socket; Device: Microprocessor-adjusting sockets

INTERVENTIONS:
Device: Static socket — For the static socket configuration, both the microprocessor control and user control are disabled, and the panels are positioned in their flush configuration to create the user's as-prescribed socket shape.
Device: User adjusted socket — Sockets are configured for user control by disabling automated control and enabling push buttons on the side of the socket to adjust socket size. Each button push effects a socket size change of approximately 0.3% volume. An upper button effects a socket size increase, and a lower button a socket size decrease. The buttons are countersunk so reduce risk of accidental pushes, and they do not function unless the user is stationary. An additional button push will not be executed until motor motion from the prior push has been completed. If a button is continuously held then the motor will continue moving until the button is released. Limits are set on cable length to ensure that sockets sizes threatening to the user's residual limb (too tight) are avoided. The push buttons effect inner-loop control that operates completely within the mechanism, achieving high-resolution adjustment of cable length with minimal error.
Device: Microprocessor-adjusting sockets — A strategy for automatically controlling the size of the socket during walking to compensate for unknown changes in limb volume will be used. The controller is essentially a regulator that continuously measures socket "fit," and adjusts the socket to maintain a prescribed reference set point. Because the fit is automatically sustained, the prosthesis user is unaware of its operation.

SUMMARY:
This is a repeated measures prospective study and is no greater than a minimal risk study. All study procedures will be conducted at the Center for the Intrepid (CFI) through collaborative efforts of the Military Performance Lab at the CFI and the Sanders lab at the University of Washington. Data collected at the CFI will be coded, compiled, and shared with the University of Washington investigators.The objective of the research is to test if microprocessor-adjusting sockets improve Service member performance in Military specific activities compared to (a) user- operated, motor-driven adjustable sockets (i.e. sockets users adjust themselves), and (b) static (traditional) sockets. Investigators also test if microprocessor-adjusting sockets better maintain socket fit and limb fluid volume, and if self-reported outcomes are more favorable than for user-operated or static sockets. The hypotheses to be tested include:

During intense Military specific tasks, compared to the user-adjusted socket and the static socket, the microprocessor-adjusting socket will:

1. minimize translational movement between the residual limb and the prosthetic socket;
2. maintain residual limb fluid volume; and
3. maximize prosthetic socket comfort.

When using the microprocessor-adjusting socket compared to the user-adjusted socket and the static socket, participants will:

1. cover the greatest distance during a simulated combat patrol;
2. perform all high intensity Military specific tasks with less pain;
3. perform a simulated combat patrol nearer to uninjured levels of performance; and
4. rank usability at a level similar to the static socket.

The specific aims are to:

1. Fabricate microprocessor-adjusting sockets specific for Service members and Veterans with goals of returning to high-level physical activities
2. Evaluate Military task performance in Service members with transtibial amputation using "Readiness Assessments," while wearing three socket configurations: microprocessor-adjusting, user-adjusting, and static

   * Simulated combat patrol in a Virtual Realty Environment
   * Military version of a Functional Capacity Evaluation
3. Characterize user preference and usability of different socket configurations

DETAILED DESCRIPTION:
The purpose of the proposed research is to evaluate the use of microprocessor-adjusting sockets during "Readiness Assessments" of Military tasks performed by Service members with transtibial amputation.

Participants will come to the Center For the Intrepid (CFI) for up to 10 visits to complete a pre-monitoring session (assess residual limb health and gather information regarding limb fluid volume); socket fitting session(s) (fitting of three sockets- static socket, a user-adjusted socket, and microprocessor-adjusting socket); and for military readiness assessments for each of the three socket conditions.

Data across the three socket conditions (static socket, user adjusted socket, and Microprocessor-adjusting sockets) will be tested for normality. When it normality can be assumed, a single factor repeated measures ANOVA will test between socket conditions. Mauchly's Test of Sphericity was be used to test if the variance is significantly different across all of the conditions. If the sphericity condition is violated, a Greenhouse-Geisser adjustment will be applied. When a significance effect is detected, pairwise comparisons using a Tukey post-hoc will be performed to determine which conditions are significantly different. When normality cannot be assumed, a Kruskal-Wallis H test will be used. When a significance effect is detected, pairwise comparisons using a Mann-Whitney post-hoc while adjusting the p-value for multiple comparisons will be performed to determine which conditions are significantly different. Statistical significance will be set to p<0.05

ELIGIBILITY:
Inclusion Criteria:

* Males and females age 18 - 55 years
* Authorized to receive care at the Center for the Intrepid
* Unilateral or bilateral transtibial amputation
* Have experience performing military relevant tasks (e.g., Active duty Service Member or Veteran)
* Current prosthesis user
* Ability to comply with instructions associated with functional testing
* Able to provide written informed consent

Exclusion Criteria:

* Self-reported inability to safely ambulate for a minimum of twenty minutes continuously and unassisted
* History of medical or psychological disease that would preclude safe gait, load carriage, physical, or cognitive functional training or testing within a virtual reality environment as determined by the provider screening the subject (i.e. moderate/severe traumatic brain injury, stroke, renal failure, cardiac or pulmonary problems disease, severe anemia, and other medical conditions)
* Any injury sustained to the upper extremity which would preclude safe physical performance testing
* Self-reported Blindness
* Self-reported Pregnancy
* Self-reported Active infection
* Weight above 250 lbs (114 kg)
* Residual limb length shorter than 9cm as this is the minimum distance necessary to attach the bio-impendence sensors
* Score greater than 20% on the Modified Oswestry Low Back Pain Questionnaire as this will indicate greater than minimal disability due to low back pain.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
Motion of the Residual Limb in the Socket | Collected during physical performance sessions (Simulated Dismounted Operations (REDoP) and Functional Capacity Evaluation-Military (FCE-M)) Approximately 3 hours.
  Angular movement between the residual limb and the prosthetic socket in the sagittal plane.
Motion of Residual Limb in the Socket | Collected during physical performance sessions (Simulated Dismounted Operations (REDoP) and Functional Capacity Evaluation-Military (FCE-M)) Approximately 3 hours.
  Translational movement between the residual limb and the prosthetic socket about the longitudinal axis of the prosthetic socket.
Self-report questionnaires of socket comfort | SCS recorded before after after each task during REDoP and FCE-M. Approximately 3 hours.
  Change in Socket Comfort Score (SCS) across the Readiness Evaluation during Simulated Dismounted Operations (REDoP) and modified Functional Capacity Evaluation-Military (FCE-M), 0-10 scale.
Readiness Evaluation during Simulated Dismounted Operations (REDoP) performance metrics | Assessment administered per condition. Approximately 55 minutes.
  Total distance traversed during REDoP assessment.
Readiness Evaluation during Simulated Dismounted Operations (REDoP) performance metrics | Recorded after each task during REDoP. Approximately 55 minutes.
  An 11-point (0-10) verbal numerical rating scale (NRS) for pain will be displayed and used to collect the individual's pain level throughout REDoP.
Functional Capacity Evaluation-Military (FCE-M) performance metrics | Assessment administered per condition. Approximately 30 minutes.
  Time to complete each sub-task of the FCE-M.
Functional Capacity Evaluation-Military (FCE-M) performance metrics | Recorded after each task during REDoP. Approximately 30 minutes.
  An 11-point (0-10) verbal numerical rating scale (NRS) for pain will be displayed and used to collect the individual's pain level throughout FCE-M.
Total score on the Post-Study System Usability Questionnaire | After each of the sessions with each socket condition, approximately 3 hours.
  This is a 19-item instrument for assessing user satisfaction with system usability. The items are 7-point graphic scales, anchored at the ends with the terms "Strongly agree" for 1, "Strongly disagree" for 7, and a "Not applicable" (N/A) point outside the scale.

SECONDARY OUTCOMES:
Readiness Evaluation during Simulated Dismounted Operations (REDoP) performance metrics | Recorded after each task during REDoP. Approximately 55 minutes.
  Marksmanship during the simulated ambushes.
Readiness Evaluation during Simulated Dismounted Operations (REDoP) performance metrics | Recorded during REDoP. Approximately 55 minutes.
  Heart rate.
Readiness Evaluation during Simulated Dismounted Operations (REDoP) performance metrics | Recorded after each task during REDoP. 5-10 sec to respond and approximately 55 minutes in total.
  Rating of perceived exertion. A standard 6-20 Borg scale will be used to collect the individual's Rating of Perceived Exertion. Subject's will be asked throughout the session to "rate the difficulty of the task" based on their fatigue level using the Borg scale.
Functional Capacity Evaluation-Military (FCE-M) performance metrics | Recorded during FCE-M. Approximately 30 minutes.
  Heart rate.
Functional Capacity Evaluation-Military (FCE-M) performance metrics | Recorded after each task during FCE-M. 5-10 sec to respond and approximately 30 minutes in total.
  Rating of perceived exertion. A standard 6-20 Borg scale will be used to collect the individual's Rating of Perceived Exertion. Subject's will be asked throughout the session to "rate the difficulty of the task" based on their fatigue level using the Borg scale.

CONTACTS AND LOCATIONS:
Overall Officials: Walter L Childers, PhD, Principal Investigator — Extremity Trauma and Amputation Center of Excellence (EACE)
Locations (1):
- Brooke Army Medical Center, Center for the Intrepid, Fort Sam Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sanders JE, Severance MR, Allyn KJ. Computer-socket manufacturing error: how much before it is clinically apparent? J Rehabil Res Dev. 2012;49(4):567-82. doi: 10.1682/jrrd.2011.05.0097. PMID 22773260
- [Background] Schnell MD BW. Management of pain in the amputee. . In: JH Bowker JM, ed. Atlas of Limb Prosthetics: Surgical, Prosthetic, and Rehabilitation Principles. 2nd ed. Chicago: Mosby-Year Book; 1982:689-706.
- [Background] Henrikson KM, Weathersby EJ, Larsen BG, Cagle JC, McLean JB, Sanders JE. An Inductive Sensing System to Measure In-Socket Residual Limb Displacements for People Using Lower-Limb Prostheses. Sensors (Basel). 2018 Nov 9;18(11):3840. doi: 10.3390/s18113840. PMID 30423932
- [Background] Sanders JE, Garbini JL, McLean JB, Hinrichs P, Predmore TJ, Brzostowski JT, Redd CB, Cagle JC. A motor-driven adjustable prosthetic socket operated using a mobile phone app: A technical note. Med Eng Phys. 2019 Jun;68:94-100. doi: 10.1016/j.medengphy.2019.04.003. Epub 2019 Apr 23. PMID 31028009
- [Background] Sanders JE, Zachariah SG, Jacobsen AK, Fergason JR. Changes in interface pressures and shear stresses over time on trans-tibial amputee subjects ambulating with prosthetic limbs: comparison of diurnal and six-month differences. J Biomech. 2005 Aug;38(8):1566-73. doi: 10.1016/j.jbiomech.2004.08.008. PMID 15958212
- [Background] Larsen BG, McLean JB, Redd CB, Brzostowski JT, Allyn KJ, Sanders JE. How do socket size adjustments during ambulation affect residual limb fluid volume? Case study results. JPO: Journal of Prosthetics and Orthotics. 2019;31(1):58-66.
- [Background] McLean JB, Redd CB, Larsen BG, Garbini JL, Brzostowski JT, Hafner BJ, Sanders JE. Socket size adjustments in people with transtibial amputation: Effects on residual limb fluid volume and limb-socket distance. Clin Biomech (Bristol). 2019 Mar;63:161-171. doi: 10.1016/j.clinbiomech.2019.02.022. Epub 2019 Mar 2. PMID 30901641
- [Background] Brzostowski JT, Larsen BG, Youngblood RT, Ciol MA, Hafner BJ, Gurrey CJ, McLean JB, Allyn KJ, Sanders JE. Adjustable sockets may improve residual limb fluid volume retention in transtibial prosthesis users. Prosthet Orthot Int. 2019 Jun;43(3):250-256. doi: 10.1177/0309364618820140. Epub 2019 Jan 10. PMID 30628522
- [Background] Fernie GR, Holliday PJ. Volume fluctuations in the residual limbs of lower limb amputees. Arch Phys Med Rehabil. 1982 Apr;63(4):162-5. PMID 7082139
- [Background] Larsen BG, Allyn KJ, Ciol MA, Sanders JE. Performance of a sensor to monitor socket fit: Comparison with practitioner clinical assessment. JPO: Journal of Prosthetics and Orthotics. 2019.
- [Background] Larsen BG, McLean JB, Allyn KJ, Brzostowski JT, Garbini JL, Sanders JE. How do transtibial residual limbs adjust to intermittent incremental socket volume changes? Prosthet Orthot Int. 2019 Oct;43(5):528-539. doi: 10.1177/0309364619864771. Epub 2019 Jul 24. PMID 31339448
- [Background] Collinger J, Grindle G, Heiner C, et al. Roadmap for future amputee care research. Care of the Combat Amputee. Washington, DC: Borden Institute, Walter Reed Army Medical Center; 2009.
- [Background] Berke GM, Fergason J, Milani JR, Hattingh J, McDowell M, Nguyen V, Reiber GE. Comparison of satisfaction with current prosthetic care in veterans and servicemembers from Vietnam and OIF/OEF conflicts with major traumatic limb loss. J Rehabil Res Dev. 2010;47(4):361-71. doi: 10.1682/jrrd.2009.12.0193. PMID 20803404
- [Background] Reiber GE, McFarland LV, Hubbard S, Maynard C, Blough DK, Gambel JM, Smith DG. Servicemembers and veterans with major traumatic limb loss from Vietnam war and OIF/OEF conflicts: survey methods, participants, and summary findings. J Rehabil Res Dev. 2010;47(4):275-97. doi: 10.1682/jrrd.2010.01.0009. PMID 20803399
- [Background] Force BIT. Dismounted Complex Blast Injury. Paper presented at: Report of the Army Dismounted Complex Blast Injury Task Force2011.
- [Background] Sanders JE, Harrison DS, Allyn KJ, Myers TR, Ciol MA, Tsai EC. How do sock ply changes affect residual-limb fluid volume in people with transtibial amputation? J Rehabil Res Dev. 2012;49(2):241-56. doi: 10.1682/jrrd.2011.02.0022. PMID 22773526
- [Background] Hinrichs P, Cagle JC, Sanders JE. A portable bioimpedance instrument for monitoring residual limb fluid volume in people with transtibial limb loss: A technical note. Med Eng Phys. 2019 Jun;68:101-107. doi: 10.1016/j.medengphy.2019.04.002. Epub 2019 Apr 22. PMID 31023596
- [Background] Sanders JE, Moehring MA, Rothlisberger TM, Phillips RH, Hartley T, Dietrich CR, Redd CB, Gardner DW, Cagle JC. A Bioimpedance Analysis Platform for Amputee Residual Limb Assessment. IEEE Trans Biomed Eng. 2016 Aug;63(8):1760-70. doi: 10.1109/TBME.2015.2502060. Epub 2015 Nov 19. PMID 26595906
- [Background] De Lorenzo A, Andreoli A, Matthie J, Withers P. Predicting body cell mass with bioimpedance by using theoretical methods: a technological review. J Appl Physiol (1985). 1997 May;82(5):1542-58. doi: 10.1152/jappl.1997.82.5.1542. PMID 9134904
- [Background] Fenech M, Jaffrin MY. Extracellular and intracellular volume variations during postural change measured by segmental and wrist-ankle bioimpedance spectroscopy. IEEE Trans Biomed Eng. 2004 Jan;51(1):166-75. doi: 10.1109/TBME.2003.820338. PMID 14723506
- [Background] Hanai T. Electrical properties of emulsions in emulsion science. Sherman PH. 1968.
- [Background] Sanders JE, Cagle JC, Allyn KJ, Harrison DS, Ciol MA. How do walking, standing, and resting influence transtibial amputee residual limb fluid volume? J Rehabil Res Dev. 2014;51(2):201-12. doi: 10.1682/JRRD.2013.04.0085. PMID 24933719
- [Background] Sanders JE, Cagle JC, Harrison DS, Myers TR, Allyn KJ. How does adding and removing liquid from socket bladders affect residual-limb fluid volume? J Rehabil Res Dev. 2013;50(6):845-60. doi: 10.1682/JRRD.2012.06.0121. PMID 24203546
- [Background] Sanders JE, Allyn KJ, Harrison DS, Myers TR, Ciol MA, Tsai EC. Preliminary investigation of residual-limb fluid volume changes within one day. J Rehabil Res Dev. 2012;49(10):1467-78. doi: 10.1682/jrrd.2011.12.0236. PMID 23516051
- [Background] Sanders JE, Harrison DS, Allyn KJ, Myers TR. Clinical utility of in-socket residual limb volume change measurement: case study results. Prosthet Orthot Int. 2009 Dec;33(4):378-90. doi: 10.3109/03093640903214067. PMID 19961297
- [Background] Sanders JE, Harrison DS, Cagle JC, Myers TR, Ciol MA, Allyn KJ. Post-doffing residual limb fluid volume change in people with trans-tibial amputation. Prosthet Orthot Int. 2012 Dec;36(4):443-9. doi: 10.1177/0309364612444752. Epub 2012 May 15. PMID 22588848
- [Background] Sanders JE, Harrison DS, Myers TR, Allyn KJ. Effects of elevated vacuum on in-socket residual limb fluid volume: case study results using bioimpedance analysis. J Rehabil Res Dev. 2011;48(10):1231-48. doi: 10.1682/jrrd.2010.11.0219. PMID 22234667
- [Background] Sanders JE, Hartley TL, Phillips RH, Ciol MA, Hafner BJ, Allyn KJ, Harrison DS. Does temporary socket removal affect residual limb fluid volume of trans-tibial amputees? Prosthet Orthot Int. 2016 Jun;40(3):320-8. doi: 10.1177/0309364614568413. Epub 2015 Feb 20. PMID 25710944
- [Background] Sanders JE, Redd CB, Cagle JC, Hafner BJ, Gardner D, Allyn KJ, Harrison DS, Ciol MA. Preliminary evaluation of a novel bladder-liner for facilitating residual limb fluid volume recovery without doffing. J Rehabil Res Dev. 2016;53(6):1107-1120. doi: 10.1682/JRRD.2014.12.0316. PMID 28355030
- [Background] Sanders JE, Youngblood RT, Hafner BJ, Ciol MA, Allyn KJ, Gardner D, Cagle JC, Redd CB, Dietrich CR. Residual limb fluid volume change and volume accommodation: Relationships to activity and self-report outcomes in people with trans-tibial amputation. Prosthet Orthot Int. 2018 Aug;42(4):415-427. doi: 10.1177/0309364617752983. Epub 2018 Feb 5. PMID 29402170
- [Background] Youngblood RT, Hafner BJ, Allyn KJ, Cagle JC, Hinrichs P, Redd C, Vamos AC, Ciol MA, Bean N, Sanders JE. Effects of activity intensity, time, and intermittent doffing on daily limb fluid volume change in people with transtibial amputation. Prosthet Orthot Int. 2019 Feb;43(1):28-38. doi: 10.1177/0309364618785729. Epub 2018 Jul 16. PMID 30010494
- [Background] Swanson EC, McLean JB, Allyn KJ, Redd CB, Sanders JE. Instrumented socket inserts for sensing interaction at the limb-socket interface. Med Eng Phys. 2018 Jan;51:111-118. doi: 10.1016/j.medengphy.2017.11.006. Epub 2017 Dec 8. PMID 29229405
- [Background] Cancio JM, Oliver RA, Yancosek KE. Functional Capacity Evaluation-Military: Program Description and Case Series. Mil Med. 2017 Jan;182(1):e1658-e1664. doi: 10.7205/MILMED-D-16-00072. PMID 28051990
- [Background] Gailey R, Kristal A, Lucarevic J, Harris S, Applegate B, Gaunaurd I. The development and internal consistency of the comprehensive lower limb amputee socket survey in active lower limb amputees. Prosthet Orthot Int. 2019 Feb;43(1):80-87. doi: 10.1177/0309364618791620. Epub 2018 Aug 10. PMID 30095355
- [Background] Venkatesh V, Morris MG, Davis GB, Davis FD. User acceptance of information technology: Toward a unified view. MIS quarterly. 2003:425-478.
- [Background] Keen SM, Kutter CJ, Niles BL, Krinsley KE. Psychometric properties of PTSD Checklist in sample of male veterans. J Rehabil Res Dev. 2008;45(3):465-74. doi: 10.1682/jrrd.2007.09.0138. PMID 18629754
- [Background] Lovell MR, Iverson GL, Collins MW, Podell K, Johnston KM, Pardini D, Pardini J, Norwig J, Maroon JC. Measurement of symptoms following sports-related concussion: reliability and normative data for the post-concussion scale. Appl Neuropsychol. 2006;13(3):166-74. doi: 10.1207/s15324826an1303_4. PMID 17361669
- [Background] Iverson GL, Gaetz M, Lovell MR, Collins MW. Relation between subjective fogginess and neuropsychological testing following concussion. J Int Neuropsychol Soc. 2004 Oct;10(6):904-6. doi: 10.1017/s1355617704106139. PMID 15637782
- [Background] Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-81. PMID 7154893
- [Background] Hanspal RS, Fisher K, Nieveen R. Prosthetic socket fit comfort score. Disabil Rehabil. 2003 Nov 18;25(22):1278-80. doi: 10.1080/09638280310001603983. PMID 14617445
- [Background] Cook KF, Dunn W, Griffith JW, Morrison MT, Tanquary J, Sabata D, Victorson D, Carey LM, Macdermid JC, Dudgeon BJ, Gershon RC. Pain assessment using the NIH Toolbox. Neurology. 2013 Mar 12;80(11 Suppl 3):S49-53. doi: 10.1212/WNL.0b013e3182872e80. PMID 23479545
- [Background] Rabago CA, Sheehan RC, Schmidtbauer KA, Vernon MC, Wilken JM. A novel assessment for Readiness Evaluation during Simulated Dismounted Operations: A reliability study. PLoS One. 2019 Dec 30;14(12):e0226386. doi: 10.1371/journal.pone.0226386. eCollection 2019. PMID 31887147
- [Background] Hill J, Timmis A. Exercise tolerance testing. BMJ. 2002 May 4;324(7345):1084-7. doi: 10.1136/bmj.324.7345.1084. No abstract available. PMID 11991917
- [Background] Hart SG, Staveland LE. Development of NASA-TLX (Task Load Index): Results of empirical and theoretical research. In: Advances in psychology. Vol 52. Elsevier; 1988:139-183.